CLINICAL TRIAL: NCT02859818
Title: Description of the Evolution of a Cohort of Adolescents With Type 1 Diabetes Following Their Participation in Therapeutic Education Program Based on Social Cognitive Theory: Socio-cognitive Profile, Physiological Behaviour of Therapeutic Adherence and Quality of Life
Acronym: ETPACAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RCAPHM15_0120
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Pediatric Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adolescents with type 1 diabetes (Other): adolescents with type 1 diabetes following their participation in therapeutic education program
  Interventions: Other: therapeutic education program

INTERVENTIONS:
Other: therapeutic education program

SUMMARY:
Introduction: Therapeutic Patient Education (TPE) is the key of the interdisciplinary management of type 1 diabetes for adolescents, favoring their adherence and improving their quality of life and metabolic control. Six pediatric diabetes teams have engaged in action research to build a regional ETP program based on social cognitive theory of Bandura, assuming that the learning strategies of theory, applied in ETP program, should strengthen self-efficacy of adolescents with type 1 diabetes, which could induce an improvement behaviors adherence, quality of life and physiological profile of participants about 6 months post-inclusion in the program.

Aims: The main objective is to describe the evolution over 6 months of self-efficacy in a cohort of adolescents with type 1 diabetes who followed a therapeutic education program based on social cognitive theory of Bandura in region PACA (ETPACAP program). Secondary objectives are to describe the evolution of 6 months of glycemic control, behavior of adherence, quality of life and other components of social cognitive theory for this population, to explore the effects of socio-cognitive profile on adherence, quality of life and glycemic control among adolescents with type 1 diabetes followed this program.

Method: A prospective multicenter cohort study of adolescents with type 1 diabetes who participated in ETPACAP program, consisting of three components:

* A quantitative component: collection and analysis of changes over 6 months of self-efficacy, adherence, quality of life and HbA1c levels (ANOVA repeated measures);
* A qualitative component: interviews with 32 participants at M0, M3 and M6 on the socio-cognitive factors according to Bandura (analysis continues theming);
* An integrative component, exploring the effects of the components of social cognitive theory on adherence, glycemic control and quality of life of adolescents with type 1 diabetes cohort.

Expected results: This research is expected to bring new knowledge about the ETP programs and the adolescent cohort studied to make an improvement and adjustment of educational sessions relevant to the needs and expectations of this population.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 11 and 17 years inclusive;
* Type 1 diabetes diagnosis confirmed by a doctor according to the diagnostic criteria;
* More than 6 months in the disease;
* Treatment with insulin for at least 6 months before the educational intervention;
* Inclusion in the program ETPACAP;
* Mastery of the French language written (elementary level)
* Fluency in speaking the French language (elementary level)
* Consent signed by the holders of parental authority and adolescents.

Exclusion Criteria:

* Pregnant women, parturient women or breastfeeding mothers (Article L.1121-5 of the Code of Public Health.)
* Persons deprived of liberty by a judicial or administrative decision, those hospitalized without consent under articles L. 3212-1 and L. 3213-1 that do not fall under the provisions of Article L. 1121-8 of the Code of Public Health

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy evaluated with the 10 items-SEDM | 6 months
  The self-efficacy will be evaluated with the 10 items-SEDM (Iannotti et al., 2006), translated into French by an adaptation process cross-cultural (linguistic validation and metrology)

SECONDARY OUTCOMES:
Adherence will be evaluated using 'the Diabetes Self-Management Profile "tool (DSMP) | 6 months
  Adherence will be evaluated using 'the Diabetes Self-Management Profile "tool (DSMP) (Schneider et al., 2007; Iannotti et al, 2006, Harris et al, 2000), translated into french through a process of adaptation-cultural (linguistic and metrological validation)
Quality of life will be assessed using the KIDSCREEN-27 | 6 months
  The quality of life will be assessed using the KIDSCREEN-27 (v 8-18 years) (Robitail et al., 2007). The KIDSCREEN is a self-administered generic questionnaire developed and validated as part of a European research project with children and adolescents (Kidscreen Group, 2006)
Glycemic control: glycated hemoglobin (HbA1c) | 6 months
  The glycated hemoglobin (HbA1c) in rising every medical visit (ISPAD, 2011)
Outcome expectations, socio-structural factors and personal goals | 6 months
  An individual semi-structured interview and audio-recorded will be led by a social health psychologist. The duration will not exceed 45 minutes. Identification of the participant in the qualitative component will link data from the interview with the collected quantitative data.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France